CLINICAL TRIAL: NCT02442141
Title: Cerebral Near-infrared Spectroscopy Monitoring in Infants During the Peri-operative Period: a Prospective Observational Cohort Study
Brief Title: Peri-operative NIRS Monitoring In Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 14-011407
Record Dates: First submitted 2015-05-05; First posted 2015-05-13 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia
Keywords: Near-Infrared Spectroscopy; Cerebral; Infants; Anesthesia; Neurodevelopmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to examine the effects of routine anesthesia on infant brain oxygen levels. The investigators do not know how anesthesia effects blood flow in the brain of infants during surgery. This study will help the investigators detect possible blood flow changes in the brain for infants undergoing anesthesia. A monitor and sensors (NIRS or near-infrared spectroscopy) which use light to measure oxygen levels in the blood will be used. Sensors will rest on the child's skin and record measurements before, during and after the surgery.

DETAILED DESCRIPTION:
Pre-operatively medical history will be collected along with baseline physiological data (Blood pressure, heart rate, date of birth, date of surgery, weight, gestational age at birth, gender, medical conditions, and medications). Given the importance of reliable blood pressure measurement- during the study, strict guidelines regarding proper blood pressure cuff placement and choice of cuff size will be followed. An upper extremity and the cuff index lines will be used to make sure that the cuff is appropriately sized. NIRS sensors will be applied pre-operatively in the operating room prior to induction of anesthesia. All NIRS values will be collected as blind values so as to not influence anesthetic management or clinical decisions.

Intra-operatively the NIRS values will be blindly recorded, physiological data and details of the anesthesia (the conduct of all clinical monitoring, including blood pressure measurements and anesthesia will not be affected in any way by this study). No additional blood pressure or other measurements will be made.

One week later the hospital record (for those infants still hospitalized) will be reviewed for evidence of new changes in neurological status (specifically seizures or other generalized or focal neurological deficits noted by the clinical team in the record and physical exam). For infants discharged home prior to one week after surgery, a phone call will be made to inquire about the occurrence of any events that required medical attention or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Less than 6 months
* Scheduled for intubation/anesthesia for clinical purposes for a surgical procedure in the Children's Hospital of Philadelphia (CHOP) Main operating room that is expected to last longer than 30 minutes

Exclusion Criteria:

* Children where application of the NIRS would be impractical: for example surgery on the head or neck.
* Children scheduled for cardiac surgery
* Children with known major cardiovascular shunting
* Children with known or suspected neurological abnormalities

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be identified from the operating room schedules or, for emergency cases the coordinating anesthetist will contact the study team.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
The incidence and range of cerebral deoxygenation during anesthesia in infants | Duration of surgery (Up to 6 hours)
  This data will be obtained by using an FDA-approved NIRS monitor. This device measures regional tissue hemoglobin saturation using combinations of spatially resolved near-infrared spectroscopy and modified Beer-Lambert law approaches, along with measure changes in tissue hemoglobin concentrations; in combination, these measurements allow changes in oxy- and deoxyhemoglobin concentrations in the tissue to be calculated. Data will be recorded prior to induction of anesthesia and throughout the procedure until the infant begins to wake or 30 after arrival to the unit, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Francis X McGowan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States